CLINICAL TRIAL: NCT06751004
Title: Effects Of Ballistic Six Exercises Versus Resistance-Band Exercises On Physical Performance Of Tennis Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0434
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Struck by Tennis Racquet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BALLISTIC SIX EXERCISES (Experimental): The Ballistic Six exercise uses resistance-band latex tube (red) and fitness balls (2-lb for one extremity training / 6-lb for dual extremity training). The 6 exercises includes; External rotation with latex tube, 90/90 external rotation with latex tube, overhead soccer throws using a fitness ball, 90/90 external rotation side-throw using a fitness ball, deceleration baseball throws using a fitness ball and baseball throws using a medicine ball
  Interventions: Other: BALLISTIC SIX EXERCISES
- RESISTANCE-BAND EXERCISES (Experimental): Week wise resistance-band training includes; 1-4 weeks: Standing Shoulder Press, Chest Fly, Triceps French Press, Biceps Curl, Rhomboid Squeeze, 5-6 weeks: Trunk Twist, Reverse Flies, Concentration Curl Scapular, Retraction, 7-8 weeks: Straight Arm Pull down, Chest Press, Triceps Kick Back, Rear Deltoid, Dead Lift
  Interventions: Other: RESISTANCE-BAND EXERCISES

INTERVENTIONS:
Other: BALLISTIC SIX EXERCISES — Ballistic six exercises will be given to group A and exercises of 3 sets of 10-20 repetitions will be completed, with each series offering 30-60 seconds of rest. The ballistic Six exercise uses resistance-band latex tube and fitness balls.
  Arms: BALLISTIC SIX EXERCISES
Other: RESISTANCE-BAND EXERCISES — Resistance-band exercises will be given to group B and the duration of training sessions will be 3 sets of 10-20 repetitions
  Arms: RESISTANCE-BAND EXERCISES

SUMMARY:
A randomized clinical trial will be conducted at Ghakhar Sports Complex,Gujranwala. Twenty eight subjects of both genders aged between 18 to 30 years will be selected who have been playing tennis for more than a year. Subjects will be randomized into two groups; Ballistic six exercises will be given to group A and exercises of 3 sets of 10-20 repetitions will be completed, with each series offering 30-60 seconds of rest. The ballistic Six exercise uses resistance-band latex tube and fitness balls. Resistance-band exercises will be given to group B and the duration of training sessions will be 3 sets of 10-20 repetitions.Assessments done will be sitting medicine ball throw test (SMBT) for shoulder strength, closed kinetic chain upper extremity stability test (CKUCEST) for agility, plate tapping test (PTT) for speed and kerlan jobe Orthopedic Clinical Score (KJOC) for shoulder function. Assessment will be done at baseline, post 8 weeks of training, at the end of 6 months. Data will be analyzed using SPSS software version 21.

DETAILED DESCRIPTION:
During regular training, players sustain injuries on a regular basis. Based on the fact that tennis isn't seen at all as a contact sport the majority of injuries are caused by overuse. A participant must perform a variety of quick, yet repeated shoulder action and repetitive motions put tension mostly on tissues with time, putting them at risk of damage. Current study will be done to compare the effects of ballistic six training versus resistance-band exercises on shoulder strength, agility, speed, and function in transitional tennis players.

A randomized clinical trial will be conducted at Ghakhar Sports Complex,Gujranwala. Twenty eight subjects of both genders aged between 18 to 30 years will be selected who have been playing tennis for more than a year. Subjects will be randomized into two groups; Ballistic six exercises will be given to group A and exercises of 3 sets of 10-20 repetitions will be completed, with each series offering 30-60 seconds of rest. The ballistic Six exercise uses resistance-band latex tube and fitness balls. Resistance-band exercises will be given to group B and the duration of training sessions will be 3 sets of 10-20 repetitions.Assessments done will be sitting medicine ball throw test (SMBT) for shoulder strength, closed kinetic chain upper extremity stability test (CKUCEST) for agility, plate tapping test (PTT) for speed and kerlan jobe Orthopedic Clinical Score (KJOC) for shoulder function. Assessment will be done at baseline, post 8 weeks of training. Data will be analyzed using SPSS software version 21. Normality of data will be checked, and tests will be applied according to normality of the data, either parametric or non-parametric test will be used (within a group or between two groups).

Key words: Agility, Ballistic Six Exercises, closed kinetic chain upper extremity stability test (CKUCEST), Fitness ball, Kerlan jobe Orthopedic Clinical score (KJOC), Plate tapping test (PTT), Resistance band exercises.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-30 years
* Participants with minimum of 1 year of tennis playing experience and normal BMI.
* Both Male and Female participants
* Participants willing to provide informed consent for participation.

Exclusion Criteria:

* Participants with less than 1 year of playing experience
* Participants who had history of bone or joint disease, musculoskeletal or painful condition (such as Carpal tunnel syndrome, Tennis elbow injury)
* History of neurological impairment, suffering from back pain for span of month
* Not willing to participate

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Sitting medicine ball throw test | Assessment will be done at baseline, post 8 weeks of training
  Sitting Medicine Ball Throw Test (SMBT) for shoulder strength
Closed kinetic chain upper extremity stability test | Assessment will be done at baseline, post 8 weeks of training
  Closed Kinetic Chain Upper Extremity Stability Test (CKUCEST) for agility
Plate tapping test | Assessment will be done at baseline, post 8 weeks of training
  Plate tapping test (PTT) for speed
Kerlan Jobe Orthopedic Clinical Score | Assessment will be done at baseline, post 8 weeks of training
  Kerlan Jobe Orthopedic Clinical Score (KJOC) for shoulder function

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, MS-DP, Principal Investigator — Riphah International University
Locations (1):
- Ghakhar Sports Complex, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No